CLINICAL TRIAL: NCT05410496
Title: A Prospective Cohort Study of Tenofovir Alafenamide Switching Therapy in Kidney or Liver Transplant Recipients with Chronic Hepatitis B Virus Infection
Brief Title: Tenofovir Alafenamide Switching Therapy in Kidney or Liver Transplant Recipients with Chronic HBV Infection
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Institute of Adherence to Medication (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF21160B
Record Dates: First submitted 2022-05-13; First posted 2022-06-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Safety Issues; Chronic Hepatitis B; Transplant Recipient
Keywords: renal function; hepatitis; patient adherence
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Patient Compliance | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAF switching therapy cohort (Experimental): A prospective single-arm cohort to evaluate the safety, drug adherence, and efficacy of TAF switching therapy in kidney or liver or transplant patients with chronic HBV infection.
  Interventions: Drug: Tenofovir Alafenamide 25 MG

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — To assess the safety, efficacy, and drug adherence improvement of TAF switching therapy in kidney or liver transplant patients with HBV infection.
  Other Names: TAF

SUMMARY:
tenofovir alafenamide (TAF) has been approved to be highly effective and safe in patients with chronic hepatitis B (CHB), therefore TAF may be a good option in kidney or liver transplant patients with chronic HBV infection. The aim of this prospective cohort study is to assess the safety, efficacy, and drug adherence improvement of TAF switching therapy in kidney or liver transplant patients with HBV infection.

DETAILED DESCRIPTION:
Life-long nucleos(t)ide analogue (NA) therapy has been recommended in patients with chronic HBV infection after organ transplantation, therefore the safety of long-term NA therapy is particularly important in transplant patients. Entecavir, tenofovir disoproxil fumarate (TDF), and tenofovir alafenamide (TAF) are recommended drugs for CHB patients in current guidelines because of their high potency in antiviral efficacy and low rate in virological resistance. However, the data of TAF therapy in transplant patients remain limited.

The potential nephrotoxicity and a decrease in bone mineral density (BMD) of TDF therapy have been reported in previous studies. TAF is a novel prodrug of tenofovir and is formulated to deliver the active metabolite to target cells more efficiently than TDF at a much lower dose, thereby reducing systemic exposure to tenofovir. In the randomized controlled trials of TDF versus TAF showed that virological and serological results were similar in both arms. However, patients in TAF arm had improved renal effects and BMD as compared to TDF. Improvement in renal function and BMD were also found in chronic hepatitis B patients who switched from TDF to TAF. Furthermore, in some retrospective studies, switching from entecavir to TAF may present a superior efficacy in HBV DNA suppression and HBsAg level reduction, and renal safety was comparable between the TAF switch group and the entecavir continuation group. Interestingly, switching from entecavir to TAF is associated with improvement of the medication adherence, which may be particularly important to patients under long-term NA therapy.

The clinical data of TAF therapy in transplant patients remain very limited, particularly in kidney transplant patients. With a high virological response rate and a low adverse effect (AE) rate in patients with CHB, TAF may be a good option for patients underwent liver or kidney transplantation.The aim of this study is to assess the safety, drug adherence, and efficacy of TAF switching therapy in kidney or liver or transplant patients with chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age
2. Chronic HBV infection under NA therapy other than TAF
3. Underwent kidney and/ or liver transplantation
4. Without clinical or pathologic evidence of moderate or severe rejection
5. Patients who are indicated for TAF switching therapy, such as concerns in virological response, biochemical response, drug compliance, or safety issues to other NAs.

Exclusion Criteria:

1. End stage renal disease (eGFR < 15 mL/min/1.73m2)
2. Co-infected with human immunodeficiency virus (HIV) or hepatitis C virus (HCV)
3. Any active malignancies
4. Pregnant or breast-feeding women
5. Known allergy to tenofovir-contained regimens

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate | week 48
  0-120 ml/min/1.73m2 (higher scores mean a better outcome)
HBV viral load | week 48
  0-8 log10 IU/mL; blood HBV DNA level (higher scores mean a worse outcome)
Drug adherence score | week 48 (higher scores mean a better outcome)
  Score 1-8; Morisky Medication Adherence Scale-8 questionnaire

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | week 144
  0-120 ml/min/1.73m2 (higher scores mean a better outcome)
HBV viral load | week 144
  0-8 log10 IU/mL; blood HBV DNA level (higher scores mean a worse outcome)
Drug adherence score | week 144 (higher scores mean a better outcome)
  Score 1-8; Morisky Medication Adherence Scale-8 questionnaire
Bone mineral density | week 144
  0-5 g/cm2; dual-energy X-ray absorptiometry (higher scores mean a better outcome)
Alanine aminotransferase | week 144
  0-150000 IU/mL; blood ALT level (higher scores mean a worse outcome)
Quantitative HBsAg | week 144
  0-10000 IU/mL; blood qHBsAg level (higher scores mean a worse outcome)
Liver fibrosis elastography | week 144
  0-30 kPa; ultrasound elastography (higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Tsai HJ, Chuang YW, Lee SW, Wu CY, Yeh HZ, Lee TY. Using the chronic kidney disease guidelines to evaluate the renal safety of tenofovir disoproxil fumarate in hepatitis B patients. Aliment Pharmacol Ther. 2018 Jun;47(12):1673-1681. doi: 10.1111/apt.14682. Epub 2018 Apr 25. PMID 29696665
- [Background] Casado JL. Renal and Bone Toxicity with the Use of Tenofovir: Understanding at the End. AIDS Rev. 2016 Apr-Jun;18(2):59-68. PMID 27230467
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Background] Lampertico P, Buti M, Fung S, Ahn SH, Chuang WL, Tak WY, Ramji A, Chen CY, Tam E, Bae H, Ma X, Flaherty JF, Gaggar A, Lau A, Liu Y, Wu G, Suri V, Tan SK, Subramanian GM, Trinh H, Yoon SK, Agarwal K, Lim YS, Chan HLY. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide in virologically suppressed patients with chronic hepatitis B: a randomised, double-blind, phase 3, multicentre non-inferiority study. Lancet Gastroenterol Hepatol. 2020 May;5(5):441-453. doi: 10.1016/S2468-1253(19)30421-2. Epub 2020 Feb 20. PMID 32087795
- [Background] Li ZB, Li L, Niu XX, Chen SH, Fu YM, Wang CY, Liu Y, Shao Q, Chen G, Ji D. Switching from entecavir to tenofovir alafenamide for chronic hepatitis B patients with low-level viraemia. Liver Int. 2021 Jun;41(6):1254-1264. doi: 10.1111/liv.14786. Epub 2021 Jan 19. PMID 33404182
- [Background] Hagiwara S, Nishida N, Ida H, Ueshima K, Minami Y, Takita M, Komeda Y, Kudo M. Switching from entecavir to tenofovir alafenamide versus maintaining entecavir for chronic hepatitis B. J Med Virol. 2019 Oct;91(10):1804-1810. doi: 10.1002/jmv.25515. Epub 2019 Jul 2. PMID 31199513
- [Background] Kumada T, Toyoda H, Tada T, Yasuda S, Miyake N, Tanaka J. Comparison of the impact of tenofovir alafenamide and entecavir on declines of hepatitis B surface antigen levels. Eur J Gastroenterol Hepatol. 2021 Feb 1;32(2):255-260. doi: 10.1097/MEG.0000000000001733. PMID 32282538
- [Background] Ogawa E, Nomura H, Nakamuta M, Furusyo N, Koyanagi T, Dohmen K, Ooho A, Satoh T, Kawano A, Kajiwara E, Takahashi K, Azuma K, Kato M, Shimoda S, Hayashi J; Kyushu University Liver Disease Study (KULDS) Group. Tenofovir alafenamide after switching from entecavir or nucleos(t)ide combination therapy for patients with chronic hepatitis B. Liver Int. 2020 Jul;40(7):1578-1589. doi: 10.1111/liv.14482. Epub 2020 Apr 30. PMID 32304611
- [Background] Uchida Y, Nakao M, Tsuji S, Uemura H, Kouyama JI, Naiki K, Motoya D, Sugawara K, Nakayama N, Imai Y, Tomiya T, Mochida S. Significance of switching of the nucleos(t)ide analog used to treat Japanese patients with chronic hepatitis B virus infection from entecavir to tenofovir alafenamide fumarate. J Med Virol. 2020 Mar;92(3):329-338. doi: 10.1002/jmv.25644. Epub 2019 Dec 9. PMID 31777965
- [Background] Rashidi-Alavijeh J, Straub K, Achterfeld A, Wedemeyer H, Willuweit K, Herzer K. Safety and efficacy of tenofovir alafenamide in liver transplant recipients: A single center experience. Transpl Infect Dis. 2021 Jun;23(3):e13522. doi: 10.1111/tid.13522. Epub 2020 Dec 22. PMID 33217163
- [Background] Sripongpun P, Mannalithara A, Kwo PY, Kim WR. Potential Benefits of Switching Liver Transplant Recipients to Tenofovir Alafenamide Prophylaxis. Clin Gastroenterol Hepatol. 2020 Mar;18(3):747-749. doi: 10.1016/j.cgh.2019.05.057. Epub 2019 Jun 11. PMID 31271737